CLINICAL TRIAL: NCT02889965
Title: The French Multiple Sclerosis Registry
Acronym: OFSEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL14_0385
Record Dates: First submitted 2016-08-22; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorders
Keywords: Multiple sclerosis; Pharmacoepidemiology; Disease modifying drugs; Neuro-myelitis optica
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Radiologically Isolated Syndromes (RIS)
- Clinically Isolated Syndromes (RIS)
- Primary progressive MS (PPMS)

SUMMARY:
OFSEP is an observational cohort of Multiple Sclerosis (MS) and related disorders set up in France. It aims to provide a major epidemiological tool on MS for the scientific community in France and abroad. This tool must help to answer a large number of questions concerning the causes and mechanisms of MS, the prognostic factors of disease progression, the effectiveness and safety of therapeutic drugs, the impact of the disease on patients and society, etc.

In December 2015, it has already included more than 54.000 patients. To achieve this goal, OFSEP's objectives are

* To maintain and develop the French cohort of patients suffering from MS or related diseases and syndromes. This means collecting standardized socio-demographic and clinical data as part of the routine medical follow-up of patients already in the cohort and recruitment of new patients.
* To supplement the existing clinical data with standardized and quality biological samples and MRI scans.
* To improve the previous data with medical/administrative data from the health insurance fund databases in particular, in order to get more information on comorbidity, treatment protocols and the medico-economic aspects of this disease.
* To use OFSEP infrastructures to facilitate the implementation of specific studies requiring the collection of additional data or specific patient monitoring processes.
* To ensure the availability of these data and samples to researchers, health care authorities and industrial players to enable analysis and thus provide answers to research questions or public health issues. This availability is only possible after scientific and regulatory evaluation of the request.
* To provide regular descriptions of the patient population in the cohort to offer statistics, targets and up-to-date information on this disease and thus enable a better approach to the personal, professional and social impacts of the illness, the effects of basic treatments and the requirements related to the follow-up of this disease in France.
* To conduct specific studies on the entire population of patients in the cohort (parent cohort) or on patient sub-groups with specific characteristics (nested cohorts). Four nested cohorts have been defined: patients with radiologically isolated syndromes, patients with clinically isolated syndromes, patients with primary progressive courses of the disease and patients with neuromyelitis optica (Devic's syndrome) spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

* RIS
* CIS
* MS according to McDonald 2010 criteria
* NMOSD and others as per NOMADMUS criteria
* No age limt
* All clinical courses
* Domiciliated in France
* Signed OFSEP informed consent

Exclusion Criteria:

NONE

-

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All MS and NMOSD patients domiciliated in France
Sampling Method: Non-Probability Sample
Enrollment: 54000 (Estimated)
Dates: Start 2011-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of cases of MS included | 6 months up to 8 years
number of patients | 6 months up to 8 years
demographic characteristics | 6 months up to 8 years
geographical distribution | 6 months up to 8 years
disease characteristics | 6 months up to 8 years
simple disease-modifying treatment description | 6 months up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Sandra VUKUSIC, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon / Hopital Neurologique Pierre Wertheimer, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gavoille A, Rollot F, Casey R, Debouverie M, Le Page E, Ciron J, De Seze J, Ruet A, Maillart E, Labauge P, Zephir H, Papeix C, Defer G, Lebrun-Frenay C, Moreau T, Laplaud DA, Berger E, Stankoff B, Clavelou P, Thouvenot E, Heinzlef O, Pelletier J, Al Khedr A, Casez O, Bourre B, Cabre P, Wahab A, Magy L, Camdessanche JP, Maurousset A, Moulin S, Ben NH, Boulos DD, Hankiewicz K, Neau JP, Pottier C, Nifle C, Rabilloud M, Subtil F, Vukusic S; Observatoire Francais de la Sclerose en Plaques (OFSEP) Investigators. Investigating the Long-term Effect of Pregnancy on the Course of Multiple Sclerosis Using Causal Inference. Neurology. 2023 Mar 21;100(12):e1296-e1308. doi: 10.1212/WNL.0000000000206774. Epub 2022 Dec 23. PMID 36564207
- [Derived] Signori A, Lorscheider J, Vukusic S, Trojano M, Iaffaldano P, Hillert J, Hyde R, Pellegrini F, Magyari M, Koch-Henriksen N, Sorensen PS, Spelman T, van der Walt A, Horakova D, Havrdova E, Girard M, Eichau S, Grand'Maison F, Gerlach O, Terzi M, Ozakbas S, Skibina O, Van Pesch V, Sa MJ, Prevost J, Alroughani R, McCombe PA, Gouider R, Mrabet S, Castillo-Trivino T, Zhu C, de Gans K, Sanchez-Menoyo JL, Yamout B, Khoury S, Sormani MP, Kalincik T, Butzkueven H; Big MS Data Network. Heterogeneity on long-term disability trajectories in patients with secondary progressive MS: a latent class analysis from Big MS Data network. J Neurol Neurosurg Psychiatry. 2023 Jan;94(1):23-30. doi: 10.1136/jnnp-2022-329987. Epub 2022 Sep 28. PMID 36171104